CLINICAL TRIAL: NCT00000998
Title: Evaluation of Escalating Doses of Intravenous Trimetrexate as Therapy for Previously Untreated Pneumocystis Carinii Pneumonia in AIDS Patients With Subsequent Comparison of Intravenous and Oral Pharmacokinetics
Brief Title: A Study of Trimetrexate in the Treatment of Pneumocystis Carinii Pneumonia (PCP) in Patients With AIDS Not Previously Treated for PCP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 018; 10994 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: Pneumonia, Pneumocystis Carinii; HIV Infections
Keywords: Trimetrexate; AIDS-Related Opportunistic Infections; Pneumonia, Pneumocystis carinii; Injections, Intravenous; Leucovorin; Dose-Response Relationship, Drug; Drug Therapy, Combination; Folic Acid Antagonists; Administration, Oral; Acquired Immunodeficiency Syndrome; Antineoplastic Agents
MeSH Terms: conditions — Pneumonia, Pneumocystis; HIV Infections; AIDS-Related Opportunistic Infections; Acquired Immunodeficiency Syndrome | interventions — trimetrexate glucuronate; Leucovorin

INTERVENTIONS:
Drug: Trimetrexate glucuronate
Drug: Leucovorin calcium

SUMMARY:
To evaluate the safety and effectiveness of trimetrexate (TMTX) given at increasing doses along with the leucovorin calcium (LCV) for treating Pneumocystis carinii pneumonia (PCP) in AIDS patients TMTX is an experimental new drug which is effective for treatment of PCP, but has been given to only a few patients. Therefore it is not certain if TMTX is better, the same as, or not as effective as conventional drugs against PCP.

DETAILED DESCRIPTION:
TMTX is an experimental new drug which is effective for treatment of PCP, but has been given to only a few patients. Therefore it is not certain if TMTX is better, the same as, or not as effective as conventional drugs against PCP.

Increasing doses of TMTX are used in combination with LCV as initial treatment for PCP in 50 AIDS patients. Doses are increased for 21 days on a once daily and then a twice daily basis. Dose escalations occur in subsequent groups of patients.

ELIGIBILITY:
Inclusion Criteria

Patient must:

* Have Pneumocystis carinii pneumonia (PCP) that has not been treated for current episode. PCP must be documented by observation of > 1 cluster of organisms in sputum, bronchial secretion, or lung tissue.
* Have clinical symptoms of respiratory disease or radiologic abnormalities.

Exclusion Criteria

* Patient cannot have significant emotional disorder.

Concurrent Medication: Excluded:

* Drugs likely to be bone marrow toxic.
* Investigational drugs.

Prior Medication: Excluded:

* Three patients in each group cannot have had zidovudine (AZT) for at least 2 months prior to administration of trimetrexate.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50
Dates: Study Completion 1989-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Masur H, Study Chair
Locations (1):
- Los Angeles County - USC Med Ctr, Los Angeles, California, United States

REFERENCES:
- [Background] Sattler FR, Allegra CJ, Verdegem TD, Akil B, Tuazon CU, Hughlett C, Ogata-Arakaki D, Feinberg J, Shelhamer J, Lane HC, et al. Trimetrexate-leucovorin dosage evaluation study for treatment of Pneumocystis carinii pneumonia. J Infect Dis. 1990 Jan;161(1):91-6. doi: 10.1093/infdis/161.1.91. PMID 2136905